CLINICAL TRIAL: NCT03131245
Title: Changes of Optic Nerve Sheath Diameter in Modified Prone Position in Craniosynostosis Children
Brief Title: Optic Nerve Sheath Diameter in Craniosynostosis
Acronym: ONSD
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, MD, PhD, Professor, Seoul National University Hospital
Other Study IDs: H1703-147-840
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Optic Nerve Sheath Diameter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Changes of optic nerve sheath diameter after position changes

DETAILED DESCRIPTION:
Changes of optic nerve sheath diameter after position changes from supine to prone position in children for craniosynostosis

ELIGIBILITY:
Inclusion Criteria:

* craniosynostosis

Exclusion Criteria:

* infection on eye area

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children for correction of craniosyostosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter | 10 minutes after prone position
  optic nerve sheath diameter measure with ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: No